CLINICAL TRIAL: NCT01598857
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Blisibimod in Addition to Methotrexate During Induction of Remission in Subjects With ANCA-Associated Small Vessel Vasculitis
Brief Title: BIANCA-SC: A Study of the Efficacy, Safety, and Tolerability of Blisibimod in Addition to Methotrexate During Induction of Remission in Subjects With ANCA-Associated Small Vessel Vasculitis
Acronym: BIANCA-SC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-VAS3321
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis
Keywords: granulomatosis with polyangiitis; microscopic polyangiitis; anti-neutrophil cytoplasmic antibodies; ANCA-associated vasculitis; Wegener Granulomatosis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Blisibimod (Experimental)
  Interventions: Drug: Blisibimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blisibimod
  Arms: Blisibimod
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerability of blisibimod when taken with methotrexate in the induction of remission in ANCA-Associated Small Vessel Vasculitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older (male or female).
2. Granulomatosis with polyangiitis (GPA, or Wegener's granulomatosis) or microscopic polyangiitis (MPA) according to the definitions of the American College of Rheumatology and Chapel Hill Consensus Conference.
3. Active GPA or MPA disease at screening.
4. Positive for either PR3-ANCA or MPO-ANCA at screening.
5. Subject willing to initiate corticosteroids and methotrexate (MTX) if not already on corticosteroids and/or MTX at baseline.
6. Clinical intention to prescribe MTX therapy for treatment of GPA or MPA.

Exclusion Criteria:

1. Diagnosed with Churg Strauss syndrome.
2. Severe GPA or MPA disease that would conventionally be treated with cyclophosphamide.
3. Nursing or pregnant.
4. Active systemic infection or deep-space infection.
5. Active hepatitis B, active hepatitis C or a documented history of HIV, hepatitis B, or hepatitis C.
6. Liver disease.
7. History of documented anti-glomerular basement membrane (GBM) disease.
8. Malignancy within the past 5 years.
9. History of active tuberculosis (TB) or history of TB infection.
10. Anemia, neutropenia, or thrombocytopenia.
11. Serum creatinine level greater than 2.5 mg/dL.
12. Prior administration of a B-cell modulating therapy other than rituximab.
13. Subject has not yet completed at least 3 months or 5 half-lives (whichever is longer) since ending other investigational study.
14. History of congenital immunodeficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Induction of clinical remission | 24 weeks
  Clinical remission includes the ability to taper corticosteroids.

SECONDARY OUTCOMES:
Time to complete remission | Various timepoints to 24 weeks
Time to treatment failure | Various timepoints to 24 weeks
Ability to taper corticosteroids | Various timepoints to 24 weeks
Change in baseline BVAS/WG score | Various timepoints to 24 weeks
Safety profile | Various timepoints to 24 weeks
Compare biomarker changes from baseline | Various timepoints to 24 weeks